CLINICAL TRIAL: NCT05225623
Title: A Community-based Adaptation of the Small Changes Behavioural Weight Loss Treatment Approach for Psoriatic Arthritis Patients With Comorbid Obesity
Brief Title: Small Changes Behavioural Weight Loss Treatment Approach for Psoriatic Arthritis Patients With Comorbid Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB21-2098
Record Dates: First submitted 2022-01-06; First posted 2022-02-04 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Psoriatic Arthritis; Obesity
Keywords: psoriatic arthritis; obesity; weight loss; behavioral intervention; small changes
MeSH Terms: conditions — Arthritis, Psoriatic; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants of the Small Changes BWLT will attend 16 2-hour group-based weekly sessions (in a virtual format using Zoom teleconferencing). Sessions will be facilitated by a senior master's level interventionist rigorously trained in the program's delivery. The empirically validated ASPIRE BWLT will be adapted for a PsA population with obesity based on the results of a qualitative study that is currently underway. After the 16 weekly sessions are complete, patients will attend bi-weekly follow-up sessions for an additional 8-weeks via Zoom. Follow-up sessions will also be group-based. In total, patients will be provided 16+8 (24) group BWLT sessions across the treatment and follow-up period.
  Participants in the control group will continue to receive their treatment as usual from the Balfour Medical Clinic and be put on a waitlist for the BWLT. This group will receive the same treatment as the intervention group after the intervention group has received treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 16-week behavioural weight loss classes
  Interventions: Behavioral: BWLT
- Waitlist Control (Other): Participants in this arm will receive their treatment as usual for Psoriatic Arthritis and receive BWLT after the intervention group.
  Interventions: Behavioral: Waitlist Control for BWLT

INTERVENTIONS:
Behavioral: BWLT — This group will attend 16 2-hour group-based weekly sessions in Small Changes BWLT in addition to their treatment at the Balfour Medical Clinic
  Arms: Intervention
Behavioral: Waitlist Control for BWLT — This group will receive treatment as usual at the Balfour Medical Clinic and put on a waitlist for the Small Changes BWLT program
  Arms: Waitlist Control

SUMMARY:
Psoriatic Arthritis (PsA) is a type of auto-immune condition that affects roughly 90,000 Canadians. Patients with PsA often experience joint pain, skin problems, and issues with mobility that negatively impact their quality of life. Compared to the general population, patients with PsA are at a higher risk of having obesity (excess body weight). Although there is no cure for PsA, medications can be helpful for symptoms, and weight loss can provide an added benefit to the effectiveness of medications.

Behavioral weight loss treatment (BWLT) is a proven way to lose weight and keep it off. BWLT usually includes individual or group sessions with a health professional to learn strategies and tools to change behaviours and thoughts in order to support weight loss. However, few studies have designed a BWLT with the unique needs of patients with PsA in mind.

Before testing new treatments for chronic disease in large, expensive studies, it is important to do smaller-scale research to make sure that a future large study will be successful. In line with this, the objective of our study is to test the feasibility of a future, large study of a BWLT for patients with PsA and obesity. In other words, our small feasibility study will investigate how convenient, reasonable, and acceptable the future study's procedures are, using a small group of people with PsA and obesity.

People who have PsA and obesity will take either a special BWLT program, or receive usual care for PsA from a community-based rheumatologist. Those in the BWLT group will complete 16 online group sessions to help them learn cognitive and behavioral changes to help improve their health and manage weight. After 24 weeks, we will determine study completion rates, examine patient satisfaction, and assess whether the BWLT was provided to people as-designed. We believe this research will help with efforts to provide more effective treatments to patients with PsA to help them lose weight and improve their quality of life through reduced pain and symptoms.

DETAILED DESCRIPTION:
Background: Psoriatic Arthritis (PsA) is an inflammatory auto-immune disorder that impacts approximately 3-in-10 patients with skin psoriasis. Compared to other rheumatologic conditions, patients with PsA are at a higher risk of having comorbid obesity (i.e., BMI ≥30 kg/m2; present in 44% of PsA cases). Treating patients with PsA and comorbid obesity presents a unique challenge due to added complications of attenuated pharmacological response to treatment, and mobility issues that impact quality of life for patients. While weight-loss is known to help alleviate symptom burden and improve quality of life in patients with PsA and comorbid obesity, few studies have investigated behavioural weight-loss treatment (BWLT) in patients with PsA to support sustained weight-loss over time.

Aims: The primary aim of the proposed trial will evaluate feasibility metrics (i.e., recruitment rate, drop-out, intervention fidelity, acceptability) of a randomized controlled clinical trial testing an adaptation of a validated "small changes"-based BWLT approach. The secondary aim is to examine differences in mean weight loss, self-reported PsA symptoms (e.g., pain, mobility) and health related quality of life (HRQOL) between patients randomized to BWLT versus patients in the control condition who receive treatment as usual (at a community-based rheumatology clinic).

Methods: The proposed study is a single center, open label parallel-group randomized control feasibility trial. Our study will control for the effect of treatment as usual in a community-based rheumatology clinic (i.e., medication and behaviour self-management). Patients will undergo baseline assessments and then will be randomized (1:1) to either the "small changes" BWLT or treatment as usual (TAU). The Small Changes BWLT is a cognitive-behavioural treatment program that was developed as an alternative to traditional behavioral therapy based on high treatment failure rates and weight regain across time - particularly in high-risk populations. Patients are provided with education on weight loss-promoting behaviour changes and encouraged to set SMALL [Self-selected, Measurable, Action-Oriented, Linked to your Life, and (Time) Limited] goals aimed at increasing self-efficacy and satisfaction, while decreasing feelings of deprivation in order to achieve sustained, long term weight loss in participants. The BWLT group will receive 16, weekly, 2-hour group-based sessions led by an undergraduate-level coach (i.e., BKin). Content covered includes nutrition, physical activity, mindfulness, cognitive restructuring, managing stress, sleep, social support, and problem-solving and is consistent with recent Canadian obesity treatment guidelines. The TAU group will received usual care from the Balfour community rheumatology clinic in Penticton, B.C. Feasibility metrics (i.e., drop-out/retention rates, patient adherence, patient-reported satisfaction with the BWLT etc.) will be assessed at the primary endpoint of 24-weeks post-randomization. Secondary outcomes (weight loss, PsA symptoms, HRQOL) will be

Impact/Future Directions: The results from the proposed study will be used to inform and develop a subsequent, adequately powered, randomized controlled efficacy trial investigating the primary outcome of weight-loss among patients with PsA and obesity who receive a BWLT, relative to TAU controls. Ultimately, the implementation of the BWLT to a community-based rheumatology clinic has potential to improve the quality of life in patients with PsA and comorbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old,
* new or previous diagnosis of symptomatic psoriatic arthritis
* BMI ≥30kg/m2),
* willing to participate in a BWLT program,
* can speak and write in English to complete surveys,
* able to participate in virtual Zoom meetings (I.e., access to a computer with email, internet and a webcam)

Exclusion Criteria:

* unstable ischemic cardiovascular disease
* severe pulmonary disease
* currently pregnant or breastfeeding
* active substance use disorder (drug or alcohol),
* currently participating in another structured weight-loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability | post-intervention (i.e., immediately following the final BWLT session at 24-weeks)
  Patients will be surveyed to asses satisfaction with the intervention in terms of: BWLT content, class duration, number of sessions, instructors, follow-up support etc.). Acceptability will be measured using a combination of Likert-style response questions and text analysis of open-field responses.
Intervention Feasibility (treatment adherence, Drop out/recruitment rates, protocol adherence) | post-intervention (i.e., immediately following the final BWLT session at 24-weeks)
  Adherence to the intervention will be determined by chart review. Referral rates of eligible patients from the AF clinic will be recorded. Drop-outs will be recorded, including reasons for study drop-out if available. The clinical supervisor (Dr. Rouleau) will evaluate the interventionists' adherence to the BWLT manual and provide feedback as needed (e.g., regarding adherence to the manual, therapeutic/process skills).

SECONDARY OUTCOMES:
Change in Weight | baseline, post-intervention (i.e., immediately following the final BWLT session at 24-weeks)
  Patients will be weighed before and after the 12 week intervention and weight loss calculated in kilograms
Change in PsA symptom burden | Baseline, post-intervention (i.e., immediately following the final BWLT session at 24-weeks)
  PsA symptoms will be assessed using the EULAR Psoriatic Arthritis Impact of Disease: PsAID12 for clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural Medicine Laboratory, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No